CLINICAL TRIAL: NCT04800900
Title: Effectiveness of Pharmaceutical Interventions in the Omission of Prescription and Desprescription of Medications in Hospitalized Patients
Brief Title: Effectiveness of Pharmaceutical Interventions in Hospitalized Patients
Acronym: INFAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Márcio Galvão Guimarães de Oliveira, Clinical Professor of Pharmacy and Evidence-based Health Care, Federal University of Bahia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 41325820
Record Dates: First submitted 2021-02-02; First posted 2021-03-16 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Safety Issues

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmaceutical intervention (Experimental): A pharmacist will analyse patient's prescription, identify if there is prescribing omission and inappropriated drug prescribed and when necessary will require to doctors
  Interventions: Other: Pharmaceutical intervention

INTERVENTIONS:
Other: Pharmaceutical intervention — A pharmacist will analyse patient's prescription, identify if there is prescribing omission and inappropriated drug prescribed and when necessary will require to doctors deprescribe or introduce or remove prescribed drugs

SUMMARY:
The presence of multimorbidities is very common among the elderly, which become major consumers of medicines. The process of prescribing medicines for the elderly should be done with caution, as the use of some medications may present more risks than benefits in this range age. Potentially inappropriate prescribing for the elderly has become a global concern for the promotion of an adequate pharmacotherapy, it becomes essential to be aware of the effectiveness and safety of medicines and the knowledge of which drugs whose risks of serious adverse reactions outweigh the benefit of your referral. In this sense, the present study has aim to evaluate the effectiveness of pharmaceutical interventions in frequency of omission of drugs with proven efficacy for cardiovascular diseases and promotion of treatment prescription inappropriate and polypharmacy. A prospective quasi experimental before and after study will be carried out in elderly patients diagnosed with cardiovascular disease admitted to the Ana Nery hospital, Salvador, Bahia, Brazil. A convenience sample will be collected, the data will be released and revised in a database built in the SPSS software and analyzed in the program statistic R and SPSS. At the end of the study, it is expected a decrease in the frequency of omission of medications and promotion of prescription drugs inappropriate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cardiovascular disease
* Discharge after 24 hours

Exclusion Criteria:

* Death

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of pharmaceutical interventions measured by proportion of accepted interventions and all interventions | The acceptance of all pharmaceutical interventions related to inappropriate prescribed drugs and omission of prescription during the hospitalization of the patient will be evaluated, through study completion, an average of 1 year

SECONDARY OUTCOMES:
Incidence of polypharmacy in elderly people with cardiovascular diseases measured by prescription containing five or more drugs | First prescription after 24 hours of admission, last prescription and discharge prescription through study completion, an average of 1 year
Incidence of omission of prescription drugs with proven efficacy for cardiovascular diseases measured by the START criteria | First prescription after 24 hours of admission, last prescription and discharge prescription through study completion, an average of 1 year
Incidence of potentially inappropriate drug prescription in elderly people with cardiovascular diseases measured by the Beers criteria | First prescription after 24 hours of admission, last prescription and discharge prescription through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ana Nery, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Gama RS, Passos LC, Amorim WW, Souza RM, Oliveira MG. Reducing Anticholinergic Burden in Hospitalised Older Adults: Analysis From the INFAR Study. Basic Clin Pharmacol Toxicol. 2026 Jan;138(1):e70160. doi: 10.1111/bcpt.70160. PMID 41345711
- [Derived] Gama RS, Passos LC, Amorim WW, Souza RM, Oliveira MG. Effectiveness of Pharmacist Interventions in Improving Medication Use in Hospitalised Older Patients Diagnosed With Cardiovascular Diseases: INFAR Before-and-After Study. J Eval Clin Pract. 2025 Jun;31(4):e70190. doi: 10.1111/jep.70190. PMID 40581959